CLINICAL TRIAL: NCT06831942
Title: Attempted Suicide Short Intervention Program for Older Adults (ASSIP-OA): An RCT and a Qualitative Evaluation of a Psychosocial Intervention for Suicidal Adults Aged 65+
Brief Title: Attempted Suicide Short Intervention Program for Older Adults (ASSIP-OA): An Evaluation of a Psychosocial Intervention for Suicidal Adults Aged 65+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-07392-01; 2023-00181 (Other Grant/Funding Number: FORTE)
Record Dates: First submitted 2025-02-05; First posted 2025-02-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-05

CONDITIONS: Suicidal Ideation; Suicide Attempt; Suicide
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted; Suicide | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ASSIP-OA (Experimental): The ASSIP-OA intervention and treatment as usual (TAU)
  Interventions: Behavioral: ASSIP-OA
- Treatment as Usual (Active Comparator): Ordinary treatment
  Interventions: Other: Treatment as Usual (TAU)

INTERVENTIONS:
Behavioral: ASSIP-OA — ASSIP-OA + TAU
  * First session. Narrative interview focusing on the background of the suicidal crisis. The patient receives a psychoeducational text to read and comment on as homework.
  * Second session. Video playback. The patient and therapist watch the video recording from session 1 together, periodically pausing the video to comment and add information.
  * Third session. Compilation of a written case conceptualization of the individual's vulnerability and triggering events that preceded the suicidal crisis.
  * Fourth session. An optional extra session to further train safety strategies.
  * Fifth session (optional). Includes one or two close relatives or other support person(s), chosen by the participant. The session focus on how safety measures learned in in ASSIP-OA can be translated into everyday life.
  * Standardized letters. therapists will send standardized letters every third month during the first year and biannually during the second year.
  Arms: ASSIP-OA
Other: Treatment as Usual (TAU) — Antidepressant medication, alone or in combination with other types of psychoactive drugs (sedatives/antipsychotics/hypnotics/mood stabilizers) constitute the cornerstone of treatment for suicidal older adults. Persons with serious depression or treatment-resistant depression may be offered electroconvulsive therapy (ECT). Some persons may receive supportive/therapeutic contacts with mental health professionals (nurses/social workers/psychologists) but no psychosocial interventions designed specifically for suicidal older adults are offered as part of ordinary treatment at the participating clinics.
  Arms: Treatment as Usual

SUMMARY:
Older adults are sorely underrepresented in suicide prevention research, despite the fact that suicide rates are higher in this age group than in any other age group in Sweden and in many countries worldwide. There are extremely few clinical intervention studies that target this age group, with to date no published studies in Europe. The overall aim is to develop and test a modified version of the Attempted Suicide Short Intervention Program (ASSIP), which the investigators will adapt specifically for older adults (65+). The original ASSIP was developed in Switzerland where it has shown an 80% decrease in risk of new suicide attempts compared to ordinary treatment. In Sweden, ASSIP is currently being tested for persons aged 18+ . The investigators now propose a randomised controlled trial (RCT) to evaluate a modification of ASSIP specifically designed to meet the needs of suicidal persons aged 65 and above, the ASSIP-Older Adult program (ASSIP-OA).

Main study questions

1. Compared to treatment as usual (TAU), will the addition of the ASSIP-OA to ordinary treatment have a preventive effect on suicide and suicide attempts within 6, 12, and 24 months following the index episode?
2. Compared to TAU, do ASSIP-OA participants show better improvement in coping skills and psychiatric symptoms a) after the last session and b) at 6-,12- and 24- month follow-up?
3. Is a brief preventive intervention (ASSIP-OA) for older adults feasible, based on its acceptability, appropriateness, deliverability and fidelity? Do participants experience side effects? Do they have fewer days of inpatient care?
4. What kind of challenges and opportunities do a) older adults and b) ASSIP-OA therapists experience in relation to implementing a brief preventive intervention like ASSIP-OA? Are the modifications that the investigators made in ASSIP-OA relevant for older adults?

ELIGIBILITY:
Inclusion Criteria:

1. Age 65 and above at time of index suicide attempt or hospitalisation for serious suicidal plans.
2. A mental health care contact during the active treatment period.
3. Capable of understanding study procedures and providing informed consent.

Exclusion Criteria:

1. Clinical diagnosis of dementia or MoCa score less than -2 standard deviations from the normative score for education and age (Borland et al., 2017). Ongoing delirium, or any other condition impeding the comprehension of the study's procedures and implications that hinder the provision of informed consent.
2. Severe ongoing psychosis, severe ongoing substance use disorder, emotionally instable personality syndrome and any other condition that would require longer specialized treatment to reduce future suicidal behaviour (e.g. DBT).
3. Terminal illness.
4. Insufficient knowledge of the Swedish language (requires interpreter).
5. Aphasia or other severe communication issue or severe hearing and/or severe visual impairment that render the intervention unfeasible despite corrective aids.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2031-06 (Estimated)

PRIMARY OUTCOMES:
New suicidal episode which includes suicide attempt or death by suicide | Follow-ups at 6, 12 and 24 months
  The primary outcome variable at 6-, 12- and 24-month follow-up is any "new suicidal episode," a composite rating that is coded "yes" in the event of a) a new suicide attempt as registered in the participant's medical record or the national hospital register or b) suicide death as registered in the national cause of death register.

SECONDARY OUTCOMES:
Severity of suicidal ideation | Secondary effect measures will be collected at baseline, immediately after the intervention (for the control group 5 weeks after baseline) and at the 6-, 12- and 24-month follow-ups.
  Columbia-Suicide Severity Rating Scale (C-SSRS) Scores range from 0-5, where higher scores indicate more severe ideation.
Depressive symptoms | Secondary effect measures will be collected at baseline, immediately after the intervention (for the control group 5 weeks after baseline) and at the 6-, 12- and 24-month follow-ups
  Montgomery-Åsberg Depression Rating Scale (MADRS) Each item yields a score of 0 to 6; the overall score thus ranges from 0 to 60. Higher MADRS score indicates more severe depression.
Anxiety | Secondary effect measures will be collected at baseline, immediately after the intervention (for the control group 5 weeks after baseline) and at the 6-, 12- and 24-month follow-ups
  Generalized Anxiety Disorder 7-item scale (GAD-7). Each item yields a score of 0 to 3; the overall score thus ranges from 0 to 21. Higher GAD-7 score indicates more severely elevated anxiety.
Coping | Secondary effect measures will be collected at baseline, immediately after the intervention (for the control group 5 weeks after baseline) and at the 6-, 12- and 24-month follow-ups
  Brief - Coping Orientation to Problems Experienced Inventory (Brief-Cope) 28 item scale 1= I haven't been doing this at all 2= A little bit 3 = A medium amount 4= I've been doing this a lot. Scores are presented for three overarching coping styles as average scores (sum of item scores divided by number of items), indicating the degree to which the respondent has been engaging in that coping style.
Health-related quality of life | Secondary effect measures will be collected at baseline, immediately after the intervention (for the control group 5 weeks after baseline) and at the 6-, 12- and 24-month follow-ups
  EQ-5D-5L . The EQ-5D-5L consists of the EQ-5D descriptive system and the EQ visual analogue scale (EQ VAS). The descriptive system comprises five dimensions: Each dimension has 5 levels: A higher 1-digit number mean a worse outcome. High scores on the EQ VAS mean a better outcome.
Health-care utilization | 12- and 24-month follow-ups.
  We will assess psychiatric inpatient hospitalizations, as well as the number and type of psychiatric healthcare contacts, based on medical records.

OTHER OUTCOMES:
Therapeutic Alliance | After the second ASSIP-OA session approx 2 weeks after of study inclusion
  Working Alliance Inventory-Short Revised (WAI-SR) measures therapeutic alliance on 12 items on a 7-point Likert scale from 1 = "never" to 7 = "always. "
Side effects | After the last ASSIP-OA session approx 5 weeks after study inclusion
  Negative Effects Questionnaire (NEQ). It contains 32 items that are scored on a five point Likert-scale (0-4) and differentiates between negative effects that are attributed to treatment and those possibly caused by other circumstances, as well as one open-ended question.
Feasibility measure Acceptability | Post intervention approx after 5 weeks
  Acceptability will be addressed in the qualitative interviews with patients post intervention.
Feasibility measure - Appropriatness | Post intervention (5-weeks) and at follow upp after 6, 12 and 24 months.
  Appropriateness is measured by Cronbach alpha and mean inter-item correlation in our questionnaires.
Feasibility measure - Deliverability | Week 1,2,3,4,5
  Deliverability is measured by examining that all components of the ASSIP- OA are provided on the 3-5 sessions without having to stress through them.
Feasibility measure - Fidelity | Week 1, 2, 3, 4, 5
  To ensure good administration of the ASSIP-OA, the investigators use: (1) training manuals with checklists for the therapists to check after each session, and (2) video recordings of randomly selected ASSIP- OA sessions (15%). They are reviewed by independent assessors using a checklist to rate the therapist's competence and adherence to the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Margda Waern, Professor, Principal Investigator — Department of Psychiatry, Institute of Neuroscience and Physiology, University of Gothenburg, Gothenburg, Sweden
Locations (2):
- Sweden (2):
  - Södra Älvsborg Hospital, Borås
  - Sahlgrenska University Hospital, Gothenburg

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared publicly, as we do not have ethical approval for individual data sharing. Any inquiries regarding access to the data should be directed to the Swedish Ethical Review Board, which oversees ethical considerations related to data access and use: registrator@etikprovning.se